CLINICAL TRIAL: NCT03555344
Title: Immediate Effect of Mantra Chikitsa on Cardiovascular Parameters in Hypertensive Patients
Brief Title: Effect of Mantra on Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Swamigal Trust for Vedic Science, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP/10164
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mantra Chikitsa (Experimental): Mantra chanting for 15 mins
  Interventions: Other: Mantra Chikitsa
- Wait list control (No Intervention): Rest for 15 Mins

INTERVENTIONS:
Other: Mantra Chikitsa — Specific Mantra were given to chants for 15 mins and resting in the impact of chants for following 15 mins.
  Other Names: Mantra therapy
  Arms: Mantra Chikitsa

SUMMARY:
Mantras are specialized energized sound or words, which are defined most important sound therapy in Vedic healing. Present study was undertaken to evaluate the immediate effect of specialized Mantra chant on cardiovascular parameters in high blood pressure patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and stable hypertension
* on regular medication

Exclusion Criteria:

* Individuals diagnosed with another lung disease,
* Have psychiatric, musculoskeletal or cardiovascular diseases,
* Being smokers
* Being pregnant

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Change from baseline to half an hour
Diastolic Blood Pressure | Change from baseline to half an hour

SECONDARY OUTCOMES:
Supine heart rate (HR) | Change from baseline to half an hour

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Director — Warwick Research Services; Ravishankar Ramanathan, Principal Investigator — Swamigal Trust for Vedic Science, India; Puneet Sharma, Study Chair — NMP Medical Research Institute
Locations (1):
- NMP Medical Research Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided